CLINICAL TRIAL: NCT01976806
Title: The Effects of Docosahexaenoic Acid on Periodontitis in Adults: A Pilot Randomized Controlled Trial
Brief Title: The Effects of DHA on Periodontitis
Acronym: DAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Center for Research Resources (NCRR) (NIH); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Kenneth Mukamal, Associate Professor of Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GM-023; UL1RR025758-02 (NIH)
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Results first posted 2014-03-24 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Periodontitis; Gingivitis; Inflammation
Keywords: Docosahexaenoic acid; DHA; Periodontitis; Gingivitis; Omega-3 fatty acid; Fish oil
MeSH Terms: conditions — Periodontitis; Gingivitis; Inflammation | interventions — Aspirin; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aspirin & Docosahexaenoic acid (Experimental): Aspirin 81 mg 1 tablet by mouth daily and Docosahexanoic acid (DHA) 500 mg 4 capsules by mouth daily (total daily dose of 2 grams DHA) for 3 months
  Interventions: Drug: Aspirin; Drug: Docosahexaenoic acid
- Aspirin & Placebo (Active Comparator): Aspirin 81 mg by mouth daily and placebo (50% corn oil/50% soybean oil) 4 capsules by mouth daily for 3 months
  Interventions: Drug: Aspirin; Drug: Placebo (for Docosahexaenoic acid)

INTERVENTIONS:
Drug: Aspirin
  Other Names: Baby Aspirin; Low Dose Aspirin
Drug: Docosahexaenoic acid
  Other Names: DHA
  Arms: Aspirin & Docosahexaenoic acid
Drug: Placebo (for Docosahexaenoic acid) — Placebo (corn/soybean oil) capsules manufactured to look identical to DHA capsules
  Other Names: 50% corn oil/50% soybean oil
  Arms: Aspirin & Placebo

SUMMARY:
The purpose of this study is to determine whether docosahexaenoic acid (DHA) is effective in the treatment of periodontitis in adults.

DETAILED DESCRIPTION:
1. The primary aim of this study is to investigate the effect of docosahexaenoic acid (DHA; 2 gm/day) plus low dose aspirin (ASA 81 mg/day)compared to ASA alone on periodontitis over three months. Our hypothesis is that DHA plus ASA will improve periodontitis as measured by objective periodontal exam, including decreased pocket depth (mm), gingival index (0-3), plaque index (0-3) and bleeding on probing (yes/no) compared to ASA alone.
2. Assess the effect of DHA and ASA exposure on markers of local inflammation, including gingival crevicular fluid (GCF) CRP, IL-1 beta and IL-6 three months after exposure to DHA plus ASA compared to ASA alone.
3. Evaluate potential mechanisms through changes in the periodontal microbial flora which may occur as a result of exposure to DHA and ASA compared to ASA alone. Our hypothesis is that there will be a substantial post therapy change in the microbial flora of dental plaques, favoring bacteria associated with a lower systemic inflammatory state.
4. Assess the effect of DHA and ASA exposure on markers of systemic inflammation, including serum C-Reactive Protein (CRP), interleukin-6 (IL-6) and vascular adhesion molecule (VCAM) compared to ASA. Our hypothesis is that there will be a decrease in serum CRP, IL-6 and VCAM three months after exposure to DHA plus ASA compared to ASA alone.
5. Assess the effect of DHA and ASA exposure on markers of systemic bone turnover, including urine N-terminal telopeptide (NTx) compared to ASA. Our hypothesis is that there will be a decrease in urine NTx three months after exposure to DHA plus ASA compared to ASA alone.

ELIGIBILITY:
Inclusion Criteria:

* age >40 years
* >20 natural teeth (excluding third molars)
* no orthodontic appliances
* periodontitis defined as >4 teeth with pocket probing depths >5 mm

Exclusion Criteria:

* pregnancy
* diabetes
* severe chronic diseases
* gastrointestinal bleeding
* uncontrolled chronic diseases
* autoimmune disorders
* conditions requiring antibiotic prophylaxis
* warfarin
* clopidogrel
* antimicrobial therapy within 30 days
* chronic use of non-steroidal anti-inflammatory drugs (other than aspirin)
* omega-3 fatty acid use within 6 months
* loose teeth
* painful teeth
* periodontal abscess
* pocket depths >10 mm in >1 tooth
* periodontal therapy within the past two years
* allergy to aspirin
* allergy to fish oil
* allergy to corn oil
* allergy to soybean oil

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Asghar Z Naqvi, MD, MPH, MNS, Principal Investigator — Beth Israel Deaconess Medical Center; Harvard Medical School; Kenneth J Mukamal, MD, MPH, MA, Study Chair — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Background] Naqvi AZ, Mu L, Hasturk H, Van Dyke TE, Mukamal KJ, Goodson JM. Impact of Docosahexaenoic Acid Therapy on Subgingival Plaque Microbiota. J Periodontol. 2017 Sep;88(9):887-895. doi: 10.1902/jop.2017.160398. Epub 2017 May 18. PMID 28517974
- [Result] Naqvi AZ, Hasturk H, Mu L, Phillips RS, Davis RB, Halem S, Campos H, Goodson JM, Van Dyke TE, Mukamal KJ. Docosahexaenoic Acid and Periodontitis in Adults: A Randomized Controlled Trial. J Dent Res. 2014 Aug;93(8):767-73. doi: 10.1177/0022034514541125. Epub 2014 Jun 26. PMID 24970858

RESULTS

PARTICIPANT FLOW:
Groups:
- Aspirin & Docosahexaenoic Acid: Aspirin 81 mg 1 tablet by mouth daily and Docosahexanoic acid (DHA) 500 mg 4 capsules by mouth daily (total daily dose of 2 grams DHA) for 3 months
  Aspirin
  Docosahexaenoic acid
- Aspirin & Placebo: Aspirin 81 mg by mouth daily and placebo (50% corn oil/50% soybean oil) 4 capsules by mouth daily for 3 months
  Aspirin
  Placebo (for Docosahexaenoic acid): Placebo (corn/soybean oil) capsules manufactured to look identical to DHA capsules
Period: Overall Study
Arm/Group | Aspirin & Docosahexaenoic Acid | Aspirin & Placebo
Started | 27 | 28
Completed | 24 | 22
Not Completed | 3 | 6
Not completed — Lost to Follow-up | 1 | 4
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Population: Includes all subjects that completed follow-up
Groups:
- Total: Total of all reporting groups
Arm/Group | Aspirin & Docosahexaenoic Acid | Aspirin & Placebo | Total
Number analyzed (Participants) | 24 | 22 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (8) | 57 (8) | 55 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 21
  Male | 13 | 12 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 8 | 15
  White | 12 | 12 | 24
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1
Smoking Status [Number; unit: participants]
  Current | 1 | 1 | 2
  Former | 7 | 6 | 13
  Never | 16 | 15 | 31
BMI (kg/m2) [Number; unit: participants]
  Normal (18.5-24.9 kg/m2) | 9 | 5 | 14
  Overweight (25-30 kg/m2) | 4 | 10 | 14
  Obese (>30 kg/m2) | 11 | 7 | 18
Hypertension [Number; unit: participants]
  Hypertension | 4 | 6 | 10
  No Hypertension | 20 | 16 | 36
Hyperlipidemia [Number; unit: participants]
  Hyperlipidemia | 5 | 4 | 9
  No Hyperlipidemia | 19 | 18 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in Pocket Depth (mm)
Description: Pocket probing depth (PD) is the depth a dental probe can be inserted into a gingival pocket at a particular site (6 sites per tooth) measured in millimeters among teeth with PD greater than or equal to 5 mm (N=533 dental sites total).
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: mm
Arm/Group | Aspirin & Docosahexaenoic Acid | Aspirin & Placebo
Number analyzed (Participants) | 24 | 22
mm | -0.71 (0.07) | -0.54 (0.07)
Statistical Analysis 1: Comparison: Aspirin & Docosahexaenoic Acid vs Aspirin & Placebo; Intent-to-treat basis with a type I error rate of 0.05. The follow-up pocket depth, was assessed in linear mixed effects models with a compound-symmetry covariance structure and age, sex, BMI, race, baseline pocket depth, baseline red blood cell (RBC) DHA level (dichotomized at median), and intervention group as fixed-effect variables; Test type: Superiority or Other; p < 0.05, Mixed Models Analysis; Compound-symmetry covariance structure with age, sex, BMI, race, baseline pocket depth, baseline RBC DHA level, and intervention group variables; Mean Difference (Net) = -0.29, Standard Error of Mean 0.13 — Mean change in pocket depth (3-month follow-up minus baseline) among dental sites with baseline pocket depths >=5 mm in the DHA intervention group versus the placebo group

2. Secondary Outcome: Change in Gingival Index (0-3)
Description: Gingival Index (GI) is a measure of gingival inflammation, which is assigned a score (0-3).
  Score Criteria:
  0: No inflammation.
  1. Mild inflammation, slight change in color, slight edema, no bleeding on probing.
  2. Moderate inflammation, moderate glazing, redness, bleeding on probing.
  3. Severe inflammation, marked redness and hypertrophy, ulceration, tendency to spontaneous bleeding.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: GI units
Arm/Group | Aspirin & Docosahexaenoic Acid | Aspirin & Placebo
Number analyzed (Participants) | 24 | 22
GI units | -0.26 (0.04) | -0.07 (0.04)

3. Secondary Outcome: Change in Plaque Index (0-3)
Description: Plaque Index (PI) is a measure of gingival inflammation as induced by bacterial plaque deposition at and under the gum line.
  Score Criteria:
  0: No plaque
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth, which can not be seen with the naked eye. But only by using disclosing solution or by using probe.
  2. Moderate accumulation of deposits within the gingival pocket, on the gingival margin and/ or adjacent tooth surface, which can be seen with the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: Plaque index units
Arm/Group | Aspirin & Docosahexaenoic Acid | Aspirin & Placebo
Number analyzed (Participants) | 24 | 22
Plaque index units | -0.10 (0.06) | 0.07 (0.07)

4. Secondary Outcome: Sites With Bleeding on Probing (Yes/no)
Description: Bleeding On Probing (BOP) is a measure of gingival inflammation and tissue destruction, which describes whether or not bleeding at the dental pocket occurred following probing.
Time Frame: 3 months
Population: Results presented at 3 months; 3-months results also compared to baseline BOP using logistic regression as described in manuscript.
Measure: Count of Units; unit: Sites
Units Other Than Participants: Sites
Arm/Group | Aspirin & Docosahexaenoic Acid | Aspirin & Placebo
Number analyzed (Participants) | 24 | 22
Number analyzed (Sites) | 271 | 261
Sites | 202 | 227

5. Secondary Outcome: Gingival Crevicular Fluid High Sensitivity C-reactive Protein
Description: Gingival crevicular fluid (GCF) is the fluid bathing the teeth under the gum line. GCF samples were analyzed for high sensitivity C-reactive protein as a measure of local gingival inflammation.
Time Frame: Baseline and 3 months
Population: Performed in all participants with baseline and 3 month visits in whom usable GCF samples could be collected.
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Aspirin & Docosahexaenoic Acid | Aspirin & Placebo
Number analyzed (Participants) | 20 | 19
ng/mL | -7.3715 (3.9244) | -3.1268 (2.0415)

6. Secondary Outcome: Gingival Crevicular Fluid Interleukin-6
Description: Gingival crevicular fluid (GCF) samples were analyzed for Interleukin-6, which is a measure of local gingival inflammation.
Time Frame: Baseline and 3 months
Population: Performed in all participants with baseline and 3 month visits in whom usable GCF samples could be collected.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Aspirin & Docosahexaenoic Acid | Aspirin & Placebo
Number analyzed (Participants) | 20 | 19
pg/mL | 0.1422 (0.5273) | -0.00226 (0.3245)

7. Secondary Outcome: Gingival Crevicular Fluid Interleukin-1 Beta
Description: Gingival crevicular fluid (GCF) samples were analyzed for Interleukin-1 beta, which is a measure of local gingival inflammation.
Time Frame: Baseline and 3 months
Population: Performed in all participants with baseline and 3 month visits in whom usable GCF samples could be collected.
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Aspirin & Docosahexaenoic Acid | Aspirin & Placebo
Number analyzed (Participants) | 20 | 19
pg/mL | 0.8775 (4.7203) | 21.5816 (8.0491)

8. Secondary Outcome: Serum High-sensitivity C-reactive Protein
Description: Serum high-sensitivity C-reactive protein is a measure of systemic inflammation.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: mg/L
Arm/Group | Aspirin & Docosahexaenoic Acid | Aspirin & Placebo
Number analyzed (Participants) | 24 | 22
mg/L | -0.3695 (0.5558) | 0.7114 (0.7223)

9. Secondary Outcome: Serum High-sensitivity Interleukin-6
Description: Serum high-sensitivity interleukin-6 is a measure of systemic inflammation.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Aspirin & Docosahexaenoic Acid | Aspirin & Placebo
Number analyzed (Participants) | 20 | 21
pg/mL | 0.3295 (0.4149) | -0.0690 (0.2633)

10. Secondary Outcome: Serum Soluble Vascular Cell Adhesion Molecule
Description: Serum soluble vascular cell adhesion molecule (VCAM) is a measure of systemic inflammation.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: ng/mL
Arm/Group | Aspirin & Docosahexaenoic Acid | Aspirin & Placebo
Number analyzed (Participants) | 20 | 21
ng/mL | 4.8829 (24.3667) | 27.9409 (19.6992)

11. Secondary Outcome: Urine N-Terminal Telopeptides
Description: Urine N-Terminal Telopeptides are a measure of systemic bone turnover.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: nM BCE
Arm/Group | Aspirin & Docosahexaenoic Acid | Aspirin & Placebo
Number analyzed (Participants) | 21 | 19
nM BCE | 103.3333 (70.5656) | 61.8421 (90.5793)

12. Other Pre Specified Outcome: Change in Red Blood Cell Membrane Docosahexaenoic Acid
Description: Red blood cell phospholipid fatty acids were measured at baseline and 3-month follow up as a measure of adherence.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Error); unit: % of total RBC FA
Arm/Group | Aspirin & Docosahexaenoic Acid | Aspirin & Placebo
Number analyzed (Participants) | 21 | 20
% of total RBC FA | 2.723 (0.3882) | -0.1776 (0.1326)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | DHA 2 gm (4 Caps) + Aspirin 81 mg (1 Tablet by Mouth Per Day) | Placebo (4 Caps) + Aspirin 81 mg (1 Tablet by Mouth Per Day)
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 7/27 | 8/28
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DHA 2 gm (4 Caps) + Aspirin 81 mg (1 Tablet by Mouth Per Day) (N=27) | Placebo (4 Caps) + Aspirin 81 mg (1 Tablet by Mouth Per Day) (N=28)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 2 (2)
Gingival bleeding while flossing (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 | 1
Fatigue (General disorders) | 2 | 1
Headache (General disorders) | 2 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1
Melena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Cavity (Infections and infestations) | 0 | 1
Verbally abusive toward staff (Psychiatric disorders) | 0 | 1
Chipped tooth (General disorders) | 1 | 0
GERD (Gastrointestinal disorders) | 0 | 1
Intermittent palpitations (Cardiac disorders) | 1 | 0
Diaphoresis (General disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No